CLINICAL TRIAL: NCT00204672
Title: The Role of GER in Exercise Triggered Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: PriCara, Unit of Ortho-McNeil, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: RAB-USA-46
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2005-09

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: Achipex

SUMMARY:
HYPOTHESIS

Gastroesophageal reflux is a major contributor to exercise-triggered asthma.

Two groups of patients will be studied: those with asthma who have difficulty with exertion, those without asthma who experience difficulty with exertion. Both groups will experience gastroesophageal reflux (GER) twice of less per week. Patients will complete a treadmill exam to determine their VO2 max. They will then undergo pH monitoring while exercising for 30 minutes at 65-70% of their VO2 max. Subjects will be given placebo or acid suppression pill for 12 weeks. At the end of 12 weeks, the subjects will repeat the exercise (30 minutes) and 24-hour pH study.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE

To determine whether patients with exercise-triggered asthma experience GER during exercise.

SECONDARY OBJECTIVES

To determine whether the exercise-induced GER within the subjects relates temporally to their exertional asthma.

To evaluate the efficacy of potent acid suppression with a proton pump inhibitor in suppressing exercise-triggered GER and asthma in these subjects.

METHODS

Population to be evaluated:

Exercise-triggered asthmatics - defined as asthmatics with exertion as their primary exacerbating factor and experiencing less than two episodes of classic gastroesophageal reflux a week.

These patients will be randomized into three different treatment groups:

1. Placebo BID
2. 20 mg Aciphex QD and placebo QPM
3. 20 mg Aciphex BID

12 patients will be studied in each group.

DATA

pH data - Data will be collected on the frequency and duration of the reflux episodes (number of episodes and the percent time the esophageal pH is less than 4.0). This will then be correlated with the respiratory symptom and changes in spirometry. A symptom index will be designed to associate the episodes of reflux and bronchospasm that occur within 5 minutes of a drop in esophageal pH.

Exercise Tolerance/Symptoms - comparisons will be made between the three groups regarding symptomatology during exercise after randomization to either placebo or differing doses of Aciphex.

Spirometry testing - done after exercise test. Comparisons between baseline and following treatment Symptoms scores - both the overall numerical grades of the patients quality of life and the number of asthmatic episodes and rescue inhaler use will be compared to baseline after the 12 week study.

STUDY DURATION

The asthma database at the University covers approximately 500 patients. A database search will be performed to identify patients suitable for recruitment. Additional recruitment, if needed, will be pursued through radio advertising. Once the study is initiated, the baseline time for therapy is 12 weeks for each patient. An estimate of the time necessary to complete the study is 15 months.

STATISTICS

Exercise triggered asthma has not been well studied with respect to its relationship to GER. This study will be considered a pilot study with 12 subjects per arm. Results from this study may be used to power a follow up study.

ELIGIBILITY:
Inclusion Criteria:

* Exercise-triggered asthmatics - defined as asthmatics with exertion as their primary exacerbating factor and experiencing less than two episodes of classic gastroesophageal reflux a week.

Exclusion Criteria:

* Exclusion criteria will be the following:

  1. Severe asthma (recent or repeated hospitalizations)
  2. Severe angina, cardiac arrhythmia's, heart failure, prior MI
  3. Respiratory illness e.g. COPD
  4. Inability to receive therapy/pH probe
  5. Pregnancy
  6. Minors, prisoners, individuals unable to give informed consent
  7. Prior upper GI surgery (gastrectomy, etc)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2000-10; Study Completion 2005-09

PRIMARY OUTCOMES:
To determine whether patients with exercise-triggered asthma experience GER during exercise.

SECONDARY OUTCOMES:
To determine whether the exercise-induced GER within the subjects relates temporally to their exertional asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn A Peterson, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States